CLINICAL TRIAL: NCT02445365
Title: Effect of Remote Ischemic Conditioning (RIC) on Inflammation and Remodelling of Extracellular Matrix Proteins in Patients With Inflammatory Bowel Diseases
Brief Title: Remote Ischemic Conditioning in Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Line Elberg Godskesen, Registrar, PhD student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S-20140133
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Colitis, Ulcerative; Gastrointestinal Diseases; Pathologic Processes; Intestinal Diseases; Inflammatory Bowel Diseases
Keywords: Ulcerative colitis; Remote ischemic conditioning
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Pathologic Processes; Intestinal Diseases; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active RIC (Experimental): Daily remote ischemic conditioning for 10 days. Remote ischemic conditioning is induced by placing a blood pressure cuff around the right or left arm. The cuff is inflated to 200 mmHg and the pressure is kept for 5 minutes. Hereafter the cuff is deflated for 5 minutes completing one cyclus. This cyclus is repeated 4 times.
  Interventions: Device: AutoRIC device
- Sham (Sham Comparator): As above with a cuff pressure of 20 mmHg
  Interventions: Device: AutoRIC device

INTERVENTIONS:
Device: AutoRIC device

SUMMARY:
Ulcerative colitis (UC) is a chronic relapsing inflammatory bowel disease (IBD). At the time of diagnosis it is not possible to predict the course of the disease, which can range from a few flares in a lifetime to uncontrollable disease leading to hospitalization, surgery and stoma. There is a continuous need to improve treatment as well as diagnostic and prognostic tools.

This study evaluates the clinical efficacy, tolerability and feasibility of remote ischemic conditioning (RIC) in patients with moderate active ulcerative colitis (UC). The investigators hypothesize that RIC beyond the well known effect on reperfusion tissue damage has a clinically relevant anti-inflammatory effect in UC. RIC constitute a repeated brief and non-harmful suppression of blood circulation in a limb. The mechanism of action of RIC is likely to involve suppressed inflammation and cell death.

Our study is a randomized clinical controlled study including 38 patients. Patients will receive RIC or sham for 10 consecutive days.

The effect of RIC on active UC is evaluated by changes patient's symptoms, endoscopy findings, and various markers in the blood, faeces and the intestinal wall.

ELIGIBILITY:
Inclusion Criteria:

* Age:≥18 years
* Verified ulcerative colitis diagnosis according to clinical, endoscopic and histological standard criteria.
* Diagnosis of ulcerative colitis established for at least 6 months
* Moderate active ulcerative colitis, total Mayo score > 6
* Endoscopic subscore activity grade ≥1
* Written informed consent

Exclusion Criteria:

* Pancolitis or acute severe ulcerative colitis requiring immediate treatment
* Need for admission due to active ulcerative colitis
* Ulcerative colitis with systemic symptoms (abdominal pain, fever > 37.5 degrees, weight loss exceeding 3 kilograms).
* Patient with anemia (Haemoglobin < 8.3 mmol/l for males and < 7.3 mmol/l for females).
* Patient with ostomy or pouch.
* The patient has had a bowel resection (except appendectomy)
* The patient has constipation and/or another known bowel condition than ulcerative colitis such as IBS.
* The patient has diabetes.
* Regular intake of acetylsalicylic acid or NSAIDs
* The patient cannot understand the information material.
* The patient has had colon cancer, dysplasia or adenomatous polyps in the colon during the recent 5 year
* The patient is in a poor general condition.
* The patient has had a food poisoning within the last three months.
* The patient is pregnant at the time of inclusion or has planned pregnancy during the period of study.
* The patient is in medical treatment with cyclosporine at the beginning of the run in period.
* Treatment for ulcerative colitis treatment has been changed within two weeks before the first day in the run in period
* The patient has commenced treatment with azathioprine, 6-mercaptopurine or methotrexate within 12 weeks before the first day in the run in period.
* The patient has commenced treatment with TNF-α inhibitors within 12 weeks before the first day of the run in period.
* The patient suffers from coeliac disease or lactose intolerance.
* Antibiotic treatment within two weeks before the first day of the run in period.
* Patient has any medical, surgical condition that excludes the use of RIC.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-05; Primary Completion 2018-02 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Change in index of clinical activity - numerical change in Mayo score including endoscopic subscore | 10 days

SECONDARY OUTCOMES:
Change in fecal calprotectin. | 10 days
Change in endoscopy - central reading according to Mayo endoscopic subscore and UCEIS | 10 days
Number of patients achieving clinical remission (Mayo score <3) | 10 days
Patient experience of repeated RIC (questionnaire, including placebo recognition). | 10 days
Change in histological score of inflammation. | 10 days
Changes in serum and mucosal cytokine profile in particular Th1/Th2/Th9/Th17/Th22. measured by FlowCytomix Multiplex. | 10 days
Changes in serum markers of inflammation (serum C-reactive protein). | 10 days
Changes in serum markers of extracellular matrix proteins (C1M, C3M, C4M, P1NP and VICM). | 10 days
Changes in serum and mucosal level of CGRP, endothelin-1, endothelin-2. | 10 days
Effect of RIC in patients with active ulcerative colitis using the Langendorff model (to document activation of a cardioprotective response). | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kjeldsen, MD, PhD, Study Chair — Odense University Hospital; Line Godskesen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark